CLINICAL TRIAL: NCT04214665
Title: A Randomized, Open-label, Balanced, Two-treatment, Four-period, Two-sequence, Single Dose, Fully Replicate, Crossover, Oral Bioequivalence Study of Alpha Lipoic Acid 600 mg HR Film Coated Tablets of Llko Ilac San. Ve Tic. A.S., Turkey and Thioctacid (Alpha Lipoic Acid) 600 mg HR Film Coated Tablets of Meda Pharma GmbH& CO .KG, Germany in 28 Healthy, Adult, Human Subjects Under Fasting Conditions.
Brief Title: To Assess the Bioequivalence of Test Oral Formulation of Alpha Lipoic Acid 600 mg HR Film Coated Tablets of Ilko Ilac San. Ve Tic. A.S. Versus Reference Thioctacid (Alpha Lipoic Acid) 600 mg HR Film Coated Tablets of Meda Pharma GmbH& CO .KG, Germany.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ilko Ilac San. ve Tic. A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 070-14-TR
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Peripheral (Sensorimotor) Diabetic Polyneuropathy
Keywords: alpha-lipoic acid; bioequivalence; replicate design
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Thioctic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test/Reference (Experimental): Single dose of test tablet in period I. Followed by single dose of reference tablet in period II. First and second dose administration will be separated by a washout period of at least 5 days.
  Interventions: Drug: Alpha Lipoic acid 600 mg HR film coated tablets
- Reference/Test (Experimental): Single dose of reference tablet in period I. Followed by single dose of test tablet in period II. First and second dose administration will be separated by a washout period of at least 5 days.
  Interventions: Drug: Alpha Lipoic acid 600 mg HR film coated tablets

INTERVENTIONS:
Drug: Alpha Lipoic acid 600 mg HR film coated tablets

SUMMARY:
To assess the bioequivalence of test oral formulation of Alpha Lipoic acid 600 mg HR film coated tablets of Ilko Ilac San. Ve Tic. A.S. versus reference Thioctacid (Alpha Lipoic acid) 600 mg HR film coated tablets of Meda Pharma GmbH& CO .KG, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Human subjects aged from 22 to 45 years (inclusive of both).
* BMI range from 18.5 to 30.0 kg/m2 inclusive with the bodyweight is::>: 45 kgs.
* Normal vital signs (Blood pressure, pulse rate, respiratory rate and body temperature).
* Normal medical and surgical history as determined by the physician or principal investigator prior to start of the study.
* Normally functioning of cardiovascular, respiratory, gastrointestinal, nervous system, musculoskeletal, vascular, genitourinary, endocrine/metabolic systems.
* Normal 12-lead electrocardiogram (ECG).
* Normal chest X-Ray (PIA view).
* Subjects able to communicate effectively.
* Willing to provide informed consent and adhere to the protocol requirements.

Exclusion Criteria:

* Contraindications or hypersensitivity to Alpha Lipoic acid or any of the excipients.
* History or presence of any disease (Gastric, renal, respiratory, cardiac, neurological etc.) according to the opinion of the physician.
* History or presence of significant alcoholism or drug abuse in the past one year.
* History or presence of significant smoking (more than 09 cigarettes or bidis/day) or consumption of tobacco products (pan, gutkha) and refusal to restrain from smoking for 48.00 hours before first period check-in until last sampling.
* History or presence of significant asthma, urticaria or other allergic reactions.
* History of difficulty in donating blood or difficulty in accessibility of veins.
* Difficulty in swallowing tablets.
* Systolic blood pressure less than 110 mm Hg or more than 139 mm Hg.
* Diastolic blood pressure less than 70mm Hg or more than 89 mm Hg.
* Pulse rate less than 60/minute or more than 1 00/minute.
* Use of any prescribed medication during last two weeks or OTC medicines or herbal medicinal products during the last one week preceding the first period check-in until completion of the study.
* Major illness during 3 months before screening.
* Subjects who have been on an unusual or abnormal diet, for whatever reason e.g. because of fasting due to religious reasons during the four weeks before screening.
* Participation in a drug research study within past 3 months.
* Donation of blood in the past 3 months before screening.
* Refusal to abstain from water for at least 01.00 hour prior to dosing and for at least 02.00 hours post dose.
* Refusal to abstain from food for at least 10.00 hours before scheduled time for dosing and for at least 04.00 hours post dose.
* Refusal to abstain from alcohol or methylxanthine-containing beverages or foods (coffee, tea, carbonated drinks, chocolate) from 48.00 hours prior to first period checkin until last sampling.
* Presence of disease markers hepatitis B & C virus & VDRL.
* HIV positive.
* Positive alcohol breath test at the time of check-in.
* Positive in the urine drugs of abuse at the time of check-in.
* Evidence of an uncooperative attitude.

Ages: 22 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-12-30 (Actual); Primary Completion 2015-01-24 (Actual); Study Completion 2015-04-21 (Actual)

PRIMARY OUTCOMES:
Cmax | pre-dose [(0.00) within 2.00 hours prior to dosing] and at 0.083, 0.167, 0.25, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50,. 3.00, 4.00, 5.00, 6.00 hours post-dose.
  Peak plasma concentration
AUC0-t | pre-dose [(0.00) within 2.00 hours prior to dosing] and at 0.083, 0.167, 0.25, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50,. 3.00, 4.00, 5.00, 6.00 hours post-dose.
  Area under the plasma concentration vs. time curve till last measured time point

SECONDARY OUTCOMES:
AUC0-∞ | pre-dose [(0.00) within 2.00 hours prior to dosing] and at 0.083, 0.167, 0.25, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50,. 3.00, 4.00, 5.00, 6.00 hours post-dose.
  Area under the plasma concentration vs. time curve extrapolated to infinity
T max | pre-dose [(0.00) within 2.00 hours prior to dosing] and at 0.083, 0.167, 0.25, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50,. 3.00, 4.00, 5.00, 6.00 hours post-dose.
  Time to achieve peak plasma concentration
t1/2 | pre-dose [(0.00) within 2.00 hours prior to dosing] and at 0.083, 0.167, 0.25, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50,. 3.00, 4.00, 5.00, 6.00 hours post-dose.
  Plasma elimination half-life
Kel | pre-dose [(0.00) within 2.00 hours prior to dosing] and at 0.083, 0.167, 0.25, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50,. 3.00, 4.00, 5.00, 6.00 hours post-dose.
  Elimination rate constant
(AUC0-inf - AUC0-t) / AUC0-inf | pre-dose [(0.00) within 2.00 hours prior to dosing] and at 0.083, 0.167, 0.25, 0.33, 0.50, 0.67, 0.83, 1.00, 1.25, 1.50, 1.75, 2.00, 2.50,. 3.00, 4.00, 5.00, 6.00 hours post-dose.
  Residual area